CLINICAL TRIAL: NCT04853498
Title: A Phase I, Open-label, Dose Escalation and Expansion Study to Evaluate the Tolerance and Pharmacokinetics of TQB3720 Tablets
Brief Title: A Study to Evaluate the Tolerance and Pharmacokinetics of TQB3720 Tablets
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3720-I-01
Record Dates: First submitted 2021-04-20; First posted 2021-04-21 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3720 tablets (Experimental): TQB3720 tablets administered orally, once daily in 28-day cycle.
  Interventions: Drug: TQB3720

INTERVENTIONS:
Drug: TQB3720 — This is an androgen receptor antagonists.

SUMMARY:
This study is conducted to investigate the pharmacokinetic and safety profiles of TQB3720 in patients with metastatic castration-resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically or cytologically confirmed prostate carcinoma. 2.Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2; Life expectancy ≥12 weeks.

  3.Testosterone levels < 50 ng/dL. 4. Has received ≥1 previous regimens for metastatic castration-resistant prostate cancer.

  5.Male subjects should agree to use an adequate method of contraception starting with signing ICF through 6 months after the last dose of study.

  6.Understood and signed an informed consent form.

Exclusion Criteria:

-1.Has symptomatic brain metastases or control of symptoms < 1 month. 2.Has other malignancies within 3 years. 3.Has used second-generation androgen receptor antagonists. 4. Abnormal liver function. 5. Abnormal renal function. 6. Has received any other investigational drug within 30 days weeks before first dose.

7. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-06-19 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Baseline up to 28 days
  MTD was defined as the dose in which more than 2 of up to 6 patients developed a DLT.

SECONDARY OUTCOMES:
Cmax | 0hour, 2hour, 4hour, 8hour, 12hour, 24hour, 36hour, 48hour, 72hour, 96hour,120hour post-dose on single dose; Hour 0 of day 8、day 15、day 22；0 hour, 2 hour, 4 hour, 8 hour, 12 hour, 24 hour post-dose on multiple dose of day 28; Hour 0 of day 42 and day 56.
  Cmax is the maximum plasma concentration of TQB3720 or metabolite(s).
Tmax | 0hour, 2hour, 4hour, 8hour, 12hour, 24hour, 36hour, 48hour, 72hour, 96hour,120hour post-dose on single dose; Hour 0 of day 8、day 15、day 22；0 hour, 2 hour, 4 hour, 8 hour, 12 hour, 24 hour post-dose on multiple dose of day 28; Hour 0 of day 42 and day 56.
  To characterize the pharmacokinetics of TQB3720 by assessment of time to reach maximum plasma concentration.
AUC0-t | 0hour, 2hour, 4hour, 8hour, 12hour, 24hour, 36hour, 48hour, 72hour, 96hour,120hour post-dose on single dose; Hour 0 of day 8、day 15、day 22；0 hour, 2 hour, 4 hour, 8 hour, 12 hour, 24 hour post-dose on multiple dose of day 28; Hour 0 of day 42 and day 56.
  To characterize the pharmacokinetics of TQB3720 by assessment of area under the plasma concentration time curve from zero to infinity.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China